CLINICAL TRIAL: NCT01319643
Title: Normal Oxygenation Maintenance in Intensive Care Unit: Randomized Controlled Trial
Brief Title: Normal Oxygenation Versus Hyperoxia in the Intensive Care Unit (ICU)
Acronym: OXYGEN-ICU
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Modena and Reggio Emilia (Other)
Responsible Party: Massimo Girardis, Università di Modena e Reggio Emilia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: OXYGEN-TIPO-1.0-30-09-2009; 2009-016506-17 (EudraCT Number)
Record Dates: First submitted 2010-08-30; First posted 2011-03-22 (Estimated); Last update posted 2011-03-22 (Estimated); Status verified 2010-08

CONDITIONS: Nervous System Diseases; Respiratory Tract Diseases; Cardiovascular Diseases; Immune System Diseases
Keywords: Oxygen; Hyperoxia; Intensive care unit; Mortality; Organ dysfunction; Postoperative care
MeSH Terms: conditions — Nervous System Diseases; Respiratory Tract Diseases; Cardiovascular Diseases; Immune System Diseases; Hyperoxia | interventions — Oxygen

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Oxygenation, rigorous normal (Experimental): Patients admitted in intensive care unit for 3 days. Administration of the lowest inspiratory fraction dose of oxygen to maintain oxygen peripheral saturation (SpO2) between 94 and 98% or an arterial partial pressure of oxygen (PaO2) between 70 and 100 mmHg. No oxygen addition administer for transports or diagnostic manoeuvres. Conventional clinical criteria for airways control and ventilation technique.
  Interventions: Drug: Oxygen
- Oxygen, free conventional (No Intervention): Patients admitted in intensive care units for 3 days. Administration of oxygen inspiratory fractions to maintain SpO2 over 97%, up to a PaO2 of 150 mmHg. Oxygen addition administer for transports or diagnostic manoeuvres. Conventional clinical criteria for airways control and ventilation technique.

INTERVENTIONS:
Drug: Oxygen — The lowest inspiratory fraction of oxygen between 21 and 100% in as a short time as possible to maintain SpO2 between 94 and 98% or PaO2 between 70 and 100 mmHg.
  Arms: Oxygenation, rigorous normal

SUMMARY:
Oxygen administration is a common practice in intensive care units, although concern is growing about oxygen toxicity. The aim of the study is to access whether a rigorous maintenance of a state of normal oxygenation in critically ill patients could obtain better outcomes, such as mortality, infections and organ failures, in comparison to conventional oxygen therapy practice.

ELIGIBILITY:
Inclusion Criteria:

* all patients admitted in a post-operative and medical intensive care unit with expected admission of at least three days. Informed consensus as soon as possible

Exclusion Criteria:

* minority
* patient discharged from ICU and successively re-admitted
* patient enrolled in other studies
* expected survival shorter than 24 hours

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 660 (Estimated)
Dates: Start 2009-12; Primary Completion 2010-11 (Estimated); Study Completion 2011-11 (Estimated)

PRIMARY OUTCOMES:
Mortality in ICU | 30 days

SECONDARY OUTCOMES:
Rate of organ dysfunctions (respiratory, circulation, renal, liver) | 30 days
Rate of nosocomial blood and respiratory infections in intensive care unit and surgery site infections in hospital. | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Massimo Girardis, PD, Principal Investigator — Università di Modena e Reggio Emilia
Locations (1):
- Terapia Intensiva Post-operatoria. Azienda Ospedaliero Universitaria Policlinico di Modena, Modena, Modena, Italy

REFERENCES:
- [Derived] Girardis M, Busani S, Damiani E, Donati A, Rinaldi L, Marudi A, Morelli A, Antonelli M, Singer M. Effect of Conservative vs Conventional Oxygen Therapy on Mortality Among Patients in an Intensive Care Unit: The Oxygen-ICU Randomized Clinical Trial. JAMA. 2016 Oct 18;316(15):1583-1589. doi: 10.1001/jama.2016.11993. PMID 27706466